CLINICAL TRIAL: NCT05623332
Title: Detecting Endometriosis inTEgrins Using teChneTium-99m Imaging Study
Brief Title: DETECT (Detecting Endometriosis inTEgrins Using teChneTium-99m Imaging Study)
Status: Enrolling by invitation | Type: Observational
Sponsor: University of Oxford (Other)
Responsible Party: Sponsor
Other Study IDs: 16073
Record Dates: First submitted 2022-08-04; First posted 2022-11-21 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Endometriosis
Keywords: non-invasive diagnosis; SPECT-CT
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Ectopic endometriosis lesions samples, endometrial samples, and endometrial flush
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Maraciclatide imaging group: Women referred to the endometriosis clinic for suspected endometriosis undergoing a maraciclatide imaging scan
  Interventions: Diagnostic Test: Maraciclatide
- Control: Control group (samples but no scan) - Women undergoing surgery for any other condition than endometriosis

INTERVENTIONS:
Diagnostic Test: Maraciclatide — Imaging marker that binds to AVB3/5 lesions
  Groups: Maraciclatide imaging group

SUMMARY:
Endometriosis is a common gynaecological disease affecting 10% of the female population due to the presence of uterus-like tissue outside of the uterus, often in the pelvis. The disease causes severe lower abdominal pain mostly during the monthly period, during or after sexual intercourse, and when emptying the bowel and bladder. Currently, imaging methods such as ultrasound are ineffective at diagnosing the most common type of endometriosis, pelvic endometriosis. Therefore, we are heavily reliant on invasive surgery to make the diagnosis.

This study aims to investigate the presence of binding proteins (integrins) in endometriotic tissue which will expand our understanding of endometriosis and could be used as a target to develop a non-invasive imaging test in the future.

Women with symptoms consistent with endometriosis, who are due to undergo surgery to diagnose endometriosis at the EndoCare Unit in Oxford, will be eligible to participate. To attempt to visualise the integrins, participants will be asked to attend 2-7 days before their surgery to undergo an imaging scan with a molecular marker that has been found to highlight integrins in other conditions. The possibility of machine learning enhancement of integrin expression will be tested. The findings on the scan will be compared to the findings at surgery. Samples during surgery of endometriosis tissues, the endometrium, and salty water that has been flushed through the uterus, will be analysed in the lab to look for differences in the amount of integrin present in women with and without endometriosis and whether factors such as the phase of the menstrual cycle or hormonal treatment effect the amount seen.

DETAILED DESCRIPTION:
This study is an open-label, exploratory research in the hospital setting.

During recruitment, women will be asked if they would like to complete a 3-5 min anonymous survey investigating their experiences and preferences of diagnostic methods and the effect the diagnostic delay of endometriosis has on fertility choices. Women will not be required to complete this to participate in the study. Women who do not wish to participate in the study will still be welcome to complete the questionnaire. They will be asked to complete a second survey revisiting the same questions after the study if their diagnosis has been confirmed. It will be clearly stated that by completing the survey consent is implied.

Once a date for the surgery is confirmed they will be booked to have their imaging scan 2-7 days before in the radiology department in Bath (Royal United Hospital) or Oxford (Churchill Hospital). On the day of the scan, they will be asked to complete a questionnaire that will provide us with information on their menstrual history, medical history, hormonal influences, and other factors that may influence the results of the scan. They will have IV maraciclatide (imaging marker) administered followed by a SPECT-CT scan(s).

As this is the first time AVB3 integrins in endometiosis lesions have been investigated using this scan, the optimum timing of the scan is unknown and additional scans (maximum 6) for the first cohort of participants will help determine the optimum timing (participants will be reimbursement accordingly). After the scan(s) they will be free to go home.

Participants will be asked to complete an 'End of Study' anonymous survey after the scan before they leave, this will evaluate their experiences of undergoing a SPECT-CT to diagnose endometriosis.

For the imaging, participants will be divided into two cohorts. Cohort 1 describes the initial research participants who assist with identifying the optimum imaging time interval following IV 99mTc-maraciclatide. Participants will undergo 1-6 imaging scans at 30 minutes, 90 minutes, 3-4 hours, 6 hours, or 18-24 hours post-administration. The timepoints the participants are allocated to will be a joint decision between the participants and research team depending on the availability of the participants, scanning slots and required timepoints. For participants in Cohort 1, the first scan will include a localization CT as part of SPECT-CT. Additional scans will include ultra-low dose CT. Depending on findings the scanning time will be refined to provide the optimal timing for visualizing lesions expressing αvβ3. The total protocol dose is 14 mSv for Cohort 1. This is equivalent to nearly 6 years of average natural background radiation in the UK. Once 4 participants with surgically confirmed endometriosis have completed each time point, the study will progress to cohort 2 using the optimum scanning. Cohort 2 describes the subsequent scans once the optimum scanning time interval has been established. One localization CT as part of SPECT will be conducted. The total protocol dose will be 9 mSv for these participants, which is equivalent to nearly 4 years of average natural background radiation in the UK. 2-7 days after participants will have their surgery as planned and if they consent they will also have samples taken for analysis of AVB3 expression.

Samples will be taken of the ectopic lesions, endometrium, and an endometrial flush (salty water flushed through the uterus). Findings on the SPECT-CT scan will be compared to laparoscopic findings to assess whether Maraciclatide can accurately detect alpha-V-beta-3 integrins in endometriotic lesions. Participants will have the opportunity to consent to their SPECT-CT images and routine ultrasound images being sent to the Oxford Applied and Theoretical Machine Learning Group. This will allow for the group to investigate whether development of machine learning algorithms can enhance the ability of alpha-V-beta-3 expression detection and other endometriosis markers.

In order to compare integrin expression in women with and without endometriosis, a control group of 25 women will be recruited to provide endometrial tissue samples and an endometrial flush sample during their planned operation. Women will be eligible to participate if they are undergoing surgery for any condition other than endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Female aged 18 years or above.
* Symptoms consistent with endometriosis and therefore due to undergo a laparoscopy for diagnostic (+/- therapeutic) purposes.
* Willing and able to comply with scheduled visits.
* In the Investigator's opinion, is able and willing to comply with all study requirements.
* Women enrolling for the tissue sample comparison group: Women undergoing planned surgery (including hysterectomy) for gynaecological disease except endometriosis e.g., fibroid-associated symptoms such as abdominal pain, abnormal uterine bleeding, fertility investigation or for laparoscopic tubal sterilisation.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the study.
* Known significant renal or hepatic impairment (E.g., eGFR <50ml/min/1.73m2 on recent blood tests).
* Any significant disease or disorder such as gynaecological cancers, in the opinion of the Investigator, may either put the participants at risk because of participation in the study or may influence the result of the study.
* High dose intravenous or intramuscular steroid in the past 12 weeks.
* Participants with a known allergy to technetium.
* Participants who have recently participated in another research study, in the opinion of the investigator will affect the results of the project.

Ages: 18 Years to 80 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Born female
Study Population: Women suspected of endometriosis due to have a diagnostic/therapeutic laparoscopy
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The correlation between locations of maraciclatide uptake identified on SPECT-CT.(described qualitatively by a radiologist) and the locations of endometriotic lesions detected during laparoscopy (described qualitatively by a surgeon) | Single comparison, maraciclatide scan to precede laparoscopy (which will occur 2-7days later)
  To assess whether alpha-v-beta-3 lesions integrins can be detected in endometriotic lesions using Maraciclatide and SPECT-CT imaging.

SECONDARY OUTCOMES:
The single best timepoint described by two radiologists following the evaluation of SPECT-CT scans at multiple time points after injection of maraciclatide. | Participants will undergo 1- 6 imaging scans at 30minutes, 90 minutes, 3-4 hours, 6 hours, or 18-24 hours post administration
  To identify the optimum imaging time interval and method following administration of intravenous maraciclatide.
The single preference of two radiologists when assessing SPECT-CT images before and after machine learning-enhancement. | Any time through the study completion, an average of 2 years
  To assess whether machine learning enhanced the ability to detect alpha-V-beta-3 integrin expression and whether this should be developed in later phase studies.
The single preference of two radiologists when assessing SPECT-CT images with and without machine learning enhancement using ultrasound scans. | All SPECT-CT images throughout study completion (average of 2 years) and any routine ultrasound images within 3 months of the scan.
  To assess whether machine learning enhanced the ability to detect alpha-V-beta-3 integrin expression and whether this should be developed in later phase studies.
The difference in alpha-V beta-3 integrin expression (using immunofluorescence) in endometrial biopsies from women with and without endometriosis. | Any time through the study completion, an average of 2 years
  To assess the angiogenic propensity of endometrial tissue in women with endometriosis.
The difference in alpha-V beta-3 integrin expression (using ELISA) in endometrial flushes from women with and without endometriosis. | Any time through the study completion, an average of 2 years
  To assess the angiogenic propensity of endometrial tissue in women with endometriosis.
The expression of alpha-V beta-3 integrin (using immunofluorescence) in the ectopic endometrial tissue samples. | Any time through the study completion, an average of 2 years
  To assess whether the phase of the cycle, hormonal influence or lesion activity affects the level of expression.
The most frequently reported highest and lowest preference for diagnostic technique presented as a percentage. | Any time through the study completion, an average of 2 years
  A national survey released via patient advocacy organisations and to those participating in the imaging study to explore the experiences and preferences of diagnostic methods in individuals undergoing investigation for endometriosis.
VAS satisfaction and acceptability rating (0 lowest - 100 highest) of participants who have undergone a SPECT-CT to detect alpha-v-beta-3 lesions in endometriotic tissue. | Any time through the study completion, an average of 2 years
  To determine whether SPECT-CT is received positively or negatively by participants undergoing investigation for endometriosis.
The number of respondents who have experienced a diagnostic delay and the number of those who think this delay has affected their life decisions. | Any time through the study completion, an average of 2 years
  To determine whether a delay in diagnosing endometriosis influences life decisions such as family planning.

CONTACTS AND LOCATIONS:
Locations (1):
- John Radcliffe Hospital, Oxford, OXON, United Kingdom

IPD SHARING:
Plan to Share IPD: No